CLINICAL TRIAL: NCT06970743
Title: A Phase 3, Open-Label, Randomized Study of BGB-16673 Compared to Investigator's Choice in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Previously Exposed to Covalent BTK Inhibitors
Brief Title: A Study of BGB-16673 Compared to Investigator's Choice in Participants With Relapsed/Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Previously Exposed to Covalent Bruton Tyrosine Kinase (BTK) Inhibitors
Acronym: CaDAnCe-303
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-303
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; SLL; BTK-targeted protein degrader
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: BGB-16673 Monotherapy (Experimental): Participants will receive BGB-16673 once daily until any of the treatment discontinuation criteria are met
  Interventions: Drug: BGB-16673
- Arm B: Investigator's Choice (Active Comparator): Participants will receive investigator's choice of bendamustine plus rituximab or high-dose methylprednisolone plus rituximab for up to six 28-day cycles.
  Participants with unequivocal disease progression confirmed by Independent Review Committee (IRC) may cross over to receive treatment with BGB-16673 at the Investigator's discretion
  Interventions: Drug: BGB-16673; Drug: Bendamustine; Drug: Rituximab; Drug: Methylprednisolone

INTERVENTIONS:
Drug: BGB-16673 — Administered orally
Drug: Bendamustine — Administered intravenously
  Arms: Arm B: Investigator's Choice
Drug: Rituximab — Administered intravenously
  Arms: Arm B: Investigator's Choice
Drug: Methylprednisolone — Administered intravenously
  Arms: Arm B: Investigator's Choice

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of BGB-16673 compared with investigator's choice (bendamustine plus rituximab or high-dose methylprednisolone plus rituximab) in participants with relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) previously exposed to covalent Bruton tyrosine kinase inhibitor(s) (cBTKi).

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia and small lymphocytic lymphoma are types of blood cancer that affects people around the world. People with CLL and SLL suffer from enlarged lymph nodes, spleen, or liver, or have symptoms like night sweats, weight loss and fever. They have shorter life expectancy compared to healthy people. There is an urgent need for new treatment to prolong life and control disease-related symptoms.

In this study, participants with R/R CLL or SLL who were previously exposed to a covalent BTKi will receive BGB-16673 or the investigator's choice of bendamustine plus rituximab or high-dose methylprednisolone plus rituximab. The main purpose of this study is to compare the length of time that participants live without their CLL or SLL worsening between those participants who receive BGB-16673 versus the investigator's choice of treatment. Approximately 150 participants will be included in this study in Mainland China and Taiwan. Participants will be randomly allocated to receive either BGB-16673 or the investigator's choice of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CLL/SLL, requiring treatment, based on 2018 international workshop on chronic lymphocytic leukemia (iwCLL) criteria.
2. Previously received treatment for CLL/SLL with a covalent BTKi.
3. Measurable disease by computer tomography/magnetic resonance imaging for patients with SLL.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. Adequate bone marrow function
6. Adequate kidney and liver function
7. Adequate blood clotting function

Exclusion Criteria:

1. Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation
2. 2. Prior autologous stem cell transplant (unless ≥ 3 months after transplant) or chimeric antigen receptor-T cell (unless ≥ 6 months after cell infusion)
3. History of severe allergic reactions or hypersensitivity to the active ingredient and excipients of study treatment (BGB-16673, bendamustine, or rituximab)
4. Current or history of central nervous system involvement
5. History of ischemic stroke or intracranial hemorrhage within 6 months before first dose of study drug
6. History of confirmed progressive multifocal leukoencephalopathy.
7. Active fungal, bacterial, and/or viral infection requiring parenteral systemic therapy
8. Clinically significant cardiovascular disease

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by IRC | Approximately 23 Months
  PFS is defined as time from the date of randomization to the date of first disease progression or death, whichever occurs first, as determined by IRC using modified 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for participants with R/R CLL and the Lugano Classification for patients with R/R SLL.

SECONDARY OUTCOMES:
PFS as Assessed by the Investigator | Approximately 12 Months
  PFS is defined as time from the date of randomization to the date of first disease progression or death, whichever occurs first, as determined by the investigator using modified 2018 iwCLL criteria for participants with CLL and the Lugano Classification for patients with R/R SLL.
Overall Survival (OS) | Approximately 21 Months
  OS is defined as time from the date of randomization to the date of death due to any cause.
Overall Response Rate (ORR) by IRC and Investigator Assessment | Approximately 23 Months
  ORR is defined as the percentage of participants with best overall response of complete response (CR), complete response with incomplete bone marrow recovery (Cri), nodular partial remission (nPR), or partial response (PR) as assessed by the IRC or by the investigator.
Rate of Partial Response with Lymphocytosis (PR-L) or Higher Determined by Investigator Assessment | Approximately 23 Months
  Rate of PR-L or higher is defined as the percentage of participants with a best overall response of complete response (CR), complete response with incomplete bone marrow recovery (Cri), nodular partial remission (nPR), partial response (PR), or partial response with lymphocytosis (PR-L) as assessed by the Investigator.
Duration of Response (DOR) by IRC and Investigator Assessment | Approximately 9 Months
  DOR is defined as the time from initial response to disease progression or death, whichever occurs first, as assessed by the IRC or by the investigator.
Time to Response (TTR) by IRC and Investigator Assessment | Approximately 6 Months
  TTR is defined as the time from randomization until initial response, as assessed by the IRC or by the investigator.
Time to Next Anti-CLL/SLL Treatment (TTNT) | Approximately 14 Months
  TTNT is defined as the time from the date of randomization to the date of next anti-CLL/SLL treatment.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Approximately 14 Months
  Safety will be assessed by monitoring and recording of all treatment emergent adverse events (AEs) and laboratory abnormalities graded by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.
Change from baseline in European Organization of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Chronic Lymphocytic Leukemia Module 17 Items (QLQ-CLL17) Symptom Burden and Physical Condition Scales | Baseline and up to approximately 23 Months
  The symptom burden and physical condition will be measured by QLQ-CLL17. EORTC QLQ-CLL17 comprises 17 items grouped into 3 multi-item scales: 1) symptom burden, 2) physical condition/fatigue, and 3) worries/fears about health and functioning. Each question is rated using a 4-point response scale ("not at all," "a little," "quite a bit," and "very much") and the recall period for all items is the past 7 days. The scores of each subscale are calculated based on the EORTC's protocol and then transformed to a 0 to 100 scale. Higher scores represent higher levels of symptom burden, physical condition/fatigue, or worries/fears about health and functioning.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Questionnaire -Core 30 (EORTC QLQ-C30) Global Health Status (GHS)/Quality of Life (QoL) and Physical Functioning Scales | Baseline and up to approximately 23 Months
  The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 =Not at all (best) to 4 =Very Much (worst) and 2 questions answered on a 7-point scale where 1 =Very poor (worst) to 7 =Excellent (best). The scores of each subscale are calculated based on the EORTC's protocol and then transformed to a 0 to 100 scale. Higher scores in GHS and functional scales indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — BeOne Medicines
Locations (64):
- China (59):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Centerhuangpu Branch, Guangzhou, Guangdong
  - Meizhou People Hospital, Meizhou, Guangdong
  - Shenzhen Nanshan Peoples Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Red Cross Hospital of Yulin City, Yulin, Guangxi
  - Guizhou Provincial Peoples Hospital, Guiyang, Guizhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical Universitynangang Branch, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technologykaiyuan Branch, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Xuchang Central Hospitalluminghu Branch, Xuchang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial Peoples Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central Peoples Hospital, Yichang, Hubei
  - The First Peoples Hospital of Changde City, Changde, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Deyangs People Hospital, Deyang, Sichuan
  - The Second Peoples Hospital of Yibin, Yibin, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciencestuanbo Branch, Tianjin, Tianjin Municipality
  - The First Peoples Hospital of Kashgar, Kashgar, Xinjiang
  - Peoples Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Peoples Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicinechengzhan, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicineqiantang Branch, Hangzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Taiwan (5):
  - Chang Bing Show Chwan Memorial Hospital, Changhua
  - China Medical University Hospital, North Dist
  - National Cheng Kung University Hospital, North Dist
  - Koo Foundation Sun Yat Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Zhongzheng Dist

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/